CLINICAL TRIAL: NCT02343822
Title: Multiple Platelet-Rich Plasma Lateral Epidondylitis Injections Versus a Single Platelet-Rich Plasma Injection in a Double-Blinded Randomized Controlled Study (PRPLE)
Brief Title: Multiple Platelet-Rich Plasma Lateral Epidondylitis Injections Versus a Single Platelet-Rich Plasma Injection
Acronym: PRPLE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN-14-2117-B
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Tennis Elbow; Lateral Epicondylitis
Keywords: PRP; Platelet Rich Plasma; Lateral Epicondylitis; Lateral Epicondylopathy; Lateral Epicondylosis; Chronic Lateral Epicondylitis; PRPLE; Multiple PRP Injections; Multiple PRP; Platelet-Rich Plasma; Tennis Elbow; Double Blinded Randomized Controlled; Multiple vs Single PRP injections; prp tennis elbow
MeSH Terms: conditions — Tennis Elbow | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Multiple PRP Injection (Experimental): 2 PRP Injections 2 months apart
  Interventions: Other: Platelet Rich Plasma Injection
- Single PRP Injection (Experimental): 1 PRP Injection and Saline Injection 2 months apart
  Interventions: Other: Platelet Rich Plasma Injection; Other: Saline Injection
- Saline Injection (Active Comparator): 2 Saline Injections 2 months apart
  Interventions: Other: Saline Injection

INTERVENTIONS:
Other: Platelet Rich Plasma Injection — Plasma component of blood rich in growth factors
  -during the injection, 5 needle fenestrations will be done to help stimulate blood flow to the area for healing
  Other Names: PRP
  Arms: Multiple PRP Injection; Single PRP Injection
Other: Saline Injection — Saline
  -during the injection, 5 needle fenestrations will be done to help stimulate blood flow to the area for healing
  Other Names: Saline
  Arms: Saline Injection; Single PRP Injection

SUMMARY:
To determine the ideal dose of PRP for lateral epicondylitis. To see if 2 PRP injections are better than a single PRP injection or a saline injection to improve function and pain in patients with lateral epicondylitis.

DETAILED DESCRIPTION:
Is there greater clinical improvement in long term pain and function when patients receive two PRP injections instead of one? This is a double-blinded randomized controlled study to determine the ideal treatment regimen for treatment of chronic lateral epicondylitis (tennis elbow). The investigators will compare pain visual analog scale (VAS) scores and functional Disabilities of Arm, Shoulder, and Hand (DASH) Questionnaire scores of patients receiving a single PRP injection and two PRP injections.

The study will be conducted at Kaiser Modesto Sports Medicine involving 532 patients who meet strict criteria for chronic lateral epicondylitis (including greater than 2 months of chronic lateral epicondylitis and failing at least one other treatment modality). Patients are randomly divided between three groups: 234 patients will receive one PRP injection, 234 will receive two, and 64 in the control group will receive a saline injection. All participants will receive concurrent home based stretching and strengthening exercises. Results are to be measured using the Visual Analog Scale (VAS) and Disabilities of Arm, Shoulder, and Hand (DASH) Questionnaire on the initial and follow-up visits of 2, 6, and 12 months. Both measures have been validated by prior studies. Successful treatment of lateral epicondylitis will be defined as a 25% reduction in visual analog score VAS and DASH scores between initial and 6 month visits. Average control and experimental groups VAS scores are expected to be 8 out of 10 with an improvement to 7 and 6 respectively in 6 months. Average control and experimental group DASH scores are expected to be 49 with an improvement to 44 and 28 respectively in 6 months.

PRP is an effective treatment in reducing pain of chronic lateral epicondylitis. This study aims to prove there is greater clinical improvement in long term pain and function when patients receive two PRP injections instead of one.

ELIGIBILITY:
Inclusion Criteria:

1. Lateral epicondylitis - diagnosed by orthopedic or sports medicine physicians / 2 separate examinations (examination at referral / confirmatory examination at time of injection)
2. Pain at the lateral epicondyle on direct palpation
3. Pain with resistive wrist extension and/or supination
4. No clinical findings at annular ligament, radiocapitellar joint, or PIN (posterior interosseous nerve syndrome)
5. No underlying bone pathology
6. Symptoms present for > 3 months
7. Visual analog score (VAS) that is >= 5/10
8. Last steroid injection > 3 months
9. Failed previous therapy (> = 4 weeks of strap, splint, cast, injection or any other accepted therapy without satisfactory pain or function)

Exclusion Criteria:

1. Age < 18 years
2. Pregnant
3. Symptomatic Carpal Tunnel syndrome on the affected side
4. History of cervical radiculopathy
5. History of Diabetes Mellitus, Rheumatoid Arthritis, hepatitis
6. Blood disorder
7. No immunocompromised patients (Human ImmunoDeficiency Virus, cancer, immunomodulator therapies)
8. Oral Nonsteroidal Antiinflammatory in the past 1 week or Steroid Drug use in the past 3 months
9. Participation in a workers' compensation program or planning to apply for the program and/or any ongoing, pending, or planned legal action as a result of elbow pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09-20 (Actual); Study Completion 2016-09-20 (Actual)

PRIMARY OUTCOMES:
Pain | 6 months
  VAS Score
Function | 6 months
  DASH Score

CONTACTS AND LOCATIONS:
Overall Officials: Wais N Arsala, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente, Modesto, California, United States

REFERENCES:
- [Background] Anitua E, Sanchez M, Nurden AT, Zalduendo M, de la Fuente M, Orive G, Azofra J, Andia I. Autologous fibrin matrices: a potential source of biological mediators that modulate tendon cell activities. J Biomed Mater Res A. 2006 May;77(2):285-93. doi: 10.1002/jbm.a.30585. PMID 16400654
- [Result] Krogh TP, Bartels EM, Ellingsen T, Stengaard-Pedersen K, Buchbinder R, Fredberg U, Bliddal H, Christensen R. Comparative effectiveness of injection therapies in lateral epicondylitis: a systematic review and network meta-analysis of randomized controlled trials. Am J Sports Med. 2013 Jun;41(6):1435-46. doi: 10.1177/0363546512458237. Epub 2012 Sep 12. PMID 22972856
- [Result] Mishra A, Pavelko T. Treatment of chronic elbow tendinosis with buffered platelet-rich plasma. Am J Sports Med. 2006 Nov;34(11):1774-8. doi: 10.1177/0363546506288850. Epub 2006 May 30. PMID 16735582
- [Result] Mishra AK, Skrepnik NV, Edwards SG, Jones GL, Sampson S, Vermillion DA, Ramsey ML, Karli DC, Rettig AC. Efficacy of platelet-rich plasma for chronic tennis elbow: a double-blind, prospective, multicenter, randomized controlled trial of 230 patients. Am J Sports Med. 2014 Feb;42(2):463-71. doi: 10.1177/0363546513494359. Epub 2013 Jul 3. PMID 23825183
- [Result] Peerbooms JC, Sluimer J, Bruijn DJ, Gosens T. Positive effect of an autologous platelet concentrate in lateral epicondylitis in a double-blind randomized controlled trial: platelet-rich plasma versus corticosteroid injection with a 1-year follow-up. Am J Sports Med. 2010 Feb;38(2):255-62. doi: 10.1177/0363546509355445. PMID 20448192
- [Result] Gosens T, Peerbooms JC, van Laar W, den Oudsten BL. Ongoing positive effect of platelet-rich plasma versus corticosteroid injection in lateral epicondylitis: a double-blind randomized controlled trial with 2-year follow-up. Am J Sports Med. 2011 Jun;39(6):1200-8. doi: 10.1177/0363546510397173. Epub 2011 Mar 21. PMID 21422467
- [Result] Arsala W, Sharpe F. Multiple Platelet-Rich Plasma Lateral Epidondylitis Injections With No Greater Positive Effect Than A Single Platelet-Rich Plasma Injection. Med&Science in Sprts&Exercise. 2012 May44(5):S82
- [Result] Kennedy JC, Willis RB. The effects of local steroid injections on tendons: a biomechanical and microscopic correlative study. Am J Sports Med. 1976 Jan-Feb;4(1):11-21. doi: 10.1177/036354657600400103. No abstract available. PMID 937623
- [Result] Taylor DW, Petrera M, Hendry M, Theodoropoulos JS. A systematic review of the use of platelet-rich plasma in sports medicine as a new treatment for tendon and ligament injuries. Clin J Sport Med. 2011 Jul;21(4):344-52. doi: 10.1097/JSM.0b013e31821d0f65. PMID 21562414